CLINICAL TRIAL: NCT01335074
Title: Temsirolimus for the Treatment of Advanced Hepatocellular Carcinoma in Patients With Intolerance to Sorafenib
Brief Title: Temsirolimus + Sorafenib in Advanced Hepatocellular Carcinoma (HCC)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Carmen Schade-Brittinger, Coordinating Center for Clinical Studies
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRHCCTS2010
Record Dates: First submitted 2011-04-12; First posted 2011-04-13 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2011-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — temsirolimus; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temsirolimus + Sorafenib (Experimental)
  Interventions: Drug: Temsirolimus + Sorafenib

INTERVENTIONS:
Drug: Temsirolimus + Sorafenib — 200mg bid Sorafenib + 15, 20 or 25 mg Temsirolimus

SUMMARY:
Sorafenib is the standard therapy for advanced liver cancer but often shows dose-limiting toxicities with the need to reduce the applied dose of the compound. As this limits the overall response rate of the therapy, a combination with temsirolimus, an inhibitor of mTOR signaling, will be investigated regarding safety and tolerability in patients with advanced liver cancer under a reduced dose of sorafenib.

DETAILED DESCRIPTION:
Inhibitors of the PI3K/Akt and mTOR signaling pathway have recently been established as novel potent anti-cancer agents for solid and hematologic malignancies. Several pre-clinical reports have shown a good anti-tumor activity in different HCC models and first reports from clinical trials in HCC promise a good efficacy in inhibiting angiogenesis and tumor cell growth. mTOR inhibition has also been shown to enhance the activity of other cytotoxic agents.

Sorafenib also interferes with tumor cell survival, proliferation and angiogenesis by inhibiting molecular pathways independent of the PI3K/Akt/mTOR signaling. We therefore expect an at least additive effect by inhibiting two parallel but independent intracellular pathways in HCC tumor cells that will prolong overall survival and time to progression.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* Patients who have a live expectancy of at least 12 weeks
* Patients with histologically or radiologically and serologically confirmed advanced HCC; documentation of original biopsy for diagnosis is acceptable if tumor tissue is unavailable
* At least one tumor lesion that can be accurately measured in at least one dimension according to RECIST and which has not been treated with local therapy (TACE, PEI, radiofrequency ablation); CT or MRI scans should be not more than 2 weeks old to be used as baseline scan
* Patients who received sorafenib at 400 mg bid with consecutive dose reduction to 200 mg bid due to intolerance, toxicity or adverse events or patients who are not eligible for full-dose first-line therapy with sorafenib, e.g. due to myocardial ischemia.
* At least a period of 4 weeks prior to baseline scan after completion of a local therapy such as surgery, radiation therapy, hepatic arterial embolization, TACE, PEI, radiofrequency ablation, cryoablation or others
* Patients who have an ECOG PS of 0, 1 or 2 or a Karnofsky Performance Status > 70 %
* Cirrhotic status of Child-Pugh class A or B; Child-Pugh status should be calculated based on clinical findings and laboratory results during the sorafenib pretreatment period
* No signs of decompensated liver cirrhosis
* White blood cells ≥ 3,000/mm³
* Neutrophils ≥ 1,500/mm³
* Platelets ≥ 100,000/mm³
* Bilirubin ≤ 3x ULN
* AST and ALT ≤ 3x ULN
* Creatinine normal
* PTT ≤ 1.5 ULN
* INT 2.0 to 3.0
* Fasting serum cholesterol ≤ 350 mg/dL
* Triglycerides ≤ 300 mg/dL
* Proteinuria ≤ 1 g in 24 h
* No history of allergic reactions to compounds similar to temsirolimus or sorafenib
* No prior thromboembolic disease
* No history of hematemesis or hemoptysis
* No other uncontrolled illness
* Women of childbearing potential must have had a negative serum or urine pregnancy test 48 h prior to the administration of the first study treatment
* Patients who give a written informed consent obtained according to local guidelines
* No other concurrent investigational drugs or anticancer agents
* No concurrent traditional Chinese or herbal medicine (e.g. sho-saiko-to, silymarine)

Exclusion Criteria:

* Patients currently receiving chemotherapy, immunotherapy or radiotherapy or who have received these with 4 weeks of study entry except for standard sorafenib therapy
* Prior use of systemic investigational agents for HCC
* Previous concurrent cancer that is distinct in primary site or histology from HCC, except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors and any cancer curatively treated > 3 years prior to entry is permitted
* Chronic treatment with steroids or another immunosuppressive agents
* A known history of HIV seropositivity
* Renal failure requiring hemo- or peritoneal dialysis
* History of cardiac disease: congestive heart failure (NYHA > 2), active coronary artery disease, cardiac arrhythmias requiring anti-arrhythmic therapy other than b-blockers or digoxin, uncontrolled hypertension; myocardial infarction more than 6 months prior to study entry is permitted
* Comedication with known strong Cyp3A4 inhibitors or Cyp3A4/5 inducers
* Active clinically serious infections (> grade 2 CTCAE v.3.0)
* Known carcinomatous meningitis or uncontrolled brain disease
* Patients with clinically significant gastrointestinal bleeding with 30 days prior to study entry or on oral anti-vitamin K medication (except low dose coumarin, i.e. INR outside the therapeutic range of 2.0 to 3.0)
* History of organ allograft
* Uncontrolled diabetes
* Impairment of gastrointestinal function of gastrointestinal disease that may significantly alter the absorption of sorafenib (e.g. ulcerative colitis, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome)
* Patients who have not recovered from surgery
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods; if barrier contraceptives are being used, these must be continued throughout the trial by both sexes
* Patients who are using other investigational agents or who had received investigational drugs < 4 weeks prior to study entry
* Patients with contraindications to sorafenib or temsirolimus treatment.
* History of noncompliance to medical regimens
* Patients unwilling or unable to comply with the protocol
* Substance abuse, medical, psychological or social conditions that may interfere with the patients participation in the study or evaluation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 12 weeks

SECONDARY OUTCOMES:
Overall response rate | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Michl, MD, Principal Investigator — Dept. of Gastroenterology; Matthias Ocker, MD, Study Director — Inst. for Surgical Research
Locations (1):
- University Hospital Giessen and Marburg, Marburg, Germany

REFERENCES:
- See also: Related Info — http://www.uni-marburg.de/fb20/chifo